CLINICAL TRIAL: NCT05307939
Title: Phase II Trial Evaluating Selective Minimal Residual Disease Directed Adjuvant Radiation in Human Papilloma Virus Associated Oropharynx Carcinoma
Brief Title: A Study on Using Cell-Free Tumor DNA (ctDNA) Testing to Decide When to StartRoutine Treatment in People With Human Papilloma Virus (HPV)- Associated Oropharynx Cancer (OPC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-434
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: HPV; Oropharynx Cancer; HPV-Related Carcinoma; HPV-Related Malignancy; HPV Positive Oropharyngeal Squamous Cell Carcinoma
Keywords: ctDNA; NavDx test; 21-434; HPV-OPC; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Costs and Cost Analysis; Radiotherapy, Intensity-Modulated; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Screening, active surveillance, and treatment (Arm A) (Experimental): Participants who meet criteria for the treatment phase (a post-operative HPV ctDNA which rose from initial undetectable to meet HPV16 ctDNA criteria and have no clinical or radiographic evidence of gross disease) will undergo delayed standard of care adjuvant radiation (50-60 Gy administered in 1.8-2 Gy fractions) based on the patient's initial pathology. Treatment will be initiated within 4 weeks of a NavDx result. Subjects will undergo FDG PET/CT simulation and standard radiation treatment planning and this FDG PET/CT will also be utilized to rule out distant metastases. Diagnostic FDG PET/CT fusion is also allowed for treatment planning and to rule out distant metastases. Non-therapeutic assessments will be completed.
  Interventions: Diagnostic Test: HPV ctDNA Assay; Diagnostic Test: MRI Studies; Behavioral: EORTC QLQ H&N 35 and C30; Behavioral: MDADI-HN; Behavioral: COST-FACIT; Radiation: Intensity-Modulated Radiation Therapy (Arm A)
- Screening and deescalated treatment (Arm B) (Experimental): Participants who meet criteria for the de-escalated treatment phase (Arm B) will undergo adjuvant radiation (30 Gy administered in 2 Gy fractions) with concurrent chemotherapy.
  They will undergo FDG PET/CT simulation and standard radiation treatment planning and this FDG PET/CT will also be utilized to rule out distant metastases. Diagnostic FDG PET/CT fusion is also allowed for treatment planning and to rule out distant metastases. Non-therapeutic assessments will be completed and the Study calendar.
  Interventions: Diagnostic Test: HPV ctDNA Assay; Diagnostic Test: MRI Studies; Behavioral: EORTC QLQ H&N 35 and C30; Behavioral: MDADI-HN; Behavioral: COST-FACIT; Combination Product: Chemoradiation (Arm B)

INTERVENTIONS:
Diagnostic Test: HPV ctDNA Assay — HPV ctDNA evaluation will be completed using NavDx which is a validated digital droplet PCR (ddPCR) assay that targets primers and hydrolysis probes to specifically detect amplicons within the E6 and E7 genes encoded by high-risk HPV strain 16, and the E7 gene for high-risk HPV strains: 18, 31, 33, and 35.
Diagnostic Test: MRI Studies — Research MRI studies will be acquired at Memorial Sloan Kettering using a fast multi-phase spoiled gradient echo sequence. A Gadolinium-based agent will be used for DCE-MRI studies.
Behavioral: EORTC QLQ H&N 35 and C30 — The EORTC QLQ H&N 35 s a validated 35-item site specific assessment tool. The module uses 7 multi-item scales to measure problems with swallowing, senses, speech, social eating and social contact. In addition, 11 single-item scales are utilized in assessing problems with teeth, mouth opening, dry mouth, sticky saliva, coughing, feeling ill, as well as use of analgesics, nutritional supplements, feeding tube and finally, weight gain and weight loss. All of the scales and single item measures range in score from 0 to 100. High scores for the Global Health Status/QoL scale represent high QoL, high scores for the functional scales represent high/healthy levels of functioning, but high scores for the symptom scales/items represent high levels of symptomatology/problems. Scoring the two instruments yields a total of 33 distinct scores and we will examine all of these scored.
  Other Names: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Module 35
Behavioral: MDADI-HN — The MDADI-HN is a questionnaire scored on a scale of 1 to 5, consisting of global, emotional, functional, and physical subscales. The MDADI-HN evaluates the effects of dysphagia on QOL.
Behavioral: COST-FACIT — Comprehensive Score for financial Toxicity or COST survey is a validated screening tool to assess objective and subjective questions about treatment-related financial distress. It is scored from 0-44, where lower composite scores reflect greater risk of financial toxicity.
  Other Names: Comprehensive Score for financial Toxicity
Radiation: Intensity-Modulated Radiation Therapy (Arm A) — 59.4-60 Gy in 1.8-2 Gy fractions: CTV_primary, Involved/Adjacent to nodal levels. 50 Gy to this volume is allowed as per MSK institutional standards in patients with clear or close margins and 2-4 involved nodes. 45-50.4 Gy in 1.8-2 Gy fractions: Dissected node positive neck: uninvolved levels that are not adjacent to positive node - Dissected node negative neck
  Arms: Screening, active surveillance, and treatment (Arm A)
Combination Product: Chemoradiation (Arm B) — 30 Gy in 2 Gy fractions: CTV_primary, CTV_node-positive neck, CTV_node-negative neck, received de-escalated postoperative chemoradiation. Adjuvant radiation will be administered as previously outlined. Concurrent chemotherapy will be administered as per standard of care. Cisplatin will be administered concurrently with radiation. For non-cisplatin candidates, carboplatin/5fu will be administered. Reasons for using carboplatin/5FU instead of cisplatin need to be charted in the medical record, but the decision belongs to the treating physician. Cisplatin may be given up to 3 days before the scheduled dates, if necessary for medical or personal reasons
  Arms: Screening and deescalated treatment (Arm B)

SUMMARY:
This study will look at whether monitoring HPV ctDNA levels is an effective way to detect cancer relapse risk in people with HPV-OPC. All participants will have recently had surgery to treat their disease, or they will be scheduled to have this surgery.

In Arm A the researchers will see whether monitoring participants' HPV ctDNA levels can safely identify patients who do not need radiation therapy (RT) after surgery and whose RT can be delayed until their HPV ctDNA levels become detectable.

In Arm B, the researchers will see whether patients who usually need 6-6.5 weeks of CRT can be selected by HPV ctDNA to receive 3 weeks of CRT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* ECOG 0-2
* HPV-16 squamous cell carcinoma of the oropharynx or HPV-16 head and neck squamous cell carcinoma of unknown primary . HPV status must be confirmed by in-situ hybridization.
* HPV ctDNA detectable by HPV digital PCR (Naveris assay) with a minimum of 50 copies/mL pre-operatively.
* Surgical resection of all gross disease with no gross disease visualized on post-operative imaging.

  o For patients with pT0 (unknown primary) evaluation for the primary should include PET/CT, direct laryngoscopy, ipsilateral tonsillectomy, and targeted biopsy. This should be followed by a neck dissection.
* Two, undetectable (<1 copy/mL) post-operative HPV ctDNA within 2-6 weeks following surgery (blood drawn at least one week apart preferred).
* A minimum of one of the following pathologic criteria: (Arm A)

  * AJCC 7 Stage: pT0N1-N2b, pT1N1, pT2N1, or ≥pT3
  * AJCC 7 ≥pN2
  * Lymphovascular invasion
  * Perineural invasion
  * Close pathologic margin (≤ 3 mm)
* Signed informed consent form by the participant or their legally authorized representative (LAR).
* A minimum of one of the following pathologic criteria (Arm B):

  * Microscopic positive margin
  * Extracapsular extension
* Signed informed consent form by the participant or their legally authorized representative (LAR).

Additional criteria for Arm B only:

* Adequate hematologic function within 30 days prior to registration, defined as follows:

  * White Blood Count (WBC) ≥ 2 K/mcL
  * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
  * Platelets ≥ 100,000 cells/mm3
  * Hemoglobin ≥ 8.0 g/dl; Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable
* Adequate renal function within 30 days prior to registration, defined as follows:

  * Serum creatinine < 1.5 mg/dl or creatinine clearance (CC) ≥ 50 ml/min determined by 24-hour collection or estimated by Cockcroft-Gault formula:
  * CCr male = [(140 - age) x (wt in kg)] divided by [(Serum Cr mg/dl) x (72)]
  * CCr female = 0.85 x (CrCl male)
* Adequate hepatic function within 30 days prior to registration, defined as follows:

  - Bilirubin < 2 mg/dl o AST or ALT < 3 x the upper limit of normal
* Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential

Exclusion Criteria:

* Metastatic disease
* Non-HPV16 genotype (i.e. HPV-18,-31, -33, -35)
* Patients who receive surgery at outside institution. Exceptions can be made for high-volume surgical centers at the discretion of the PI/co-PI
* Prior head and neck radiation
* Patients without pre-operative HPV ctDNA or pre-operative HPV ctDNA ≤ 50 copies/mL
* Subjects with simultaneous primary cancers outside of the oropharynx

  o Note: Exceptions can be made for patients with simultaneous primaries outside of the oropharynx if determined by the PI/Co-PI, then the patient can proceed with protocol activities
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for 3 years or if cure rate from treatment at 5 years is 90% or greater

  o Note: Exceptions can be made for patients with prior invasive malignancy if determined by the PI/Co-PI, then the patient can proceed with protocol activities
* Prior systemic chemotherapy for the study cancer

  o Note: prior chemotherapy for a different cancer is allowable
* Severe, active co-morbidity defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization within 30 days of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
* Lack of ability to understand and willingness to sign a written informed consent and complete questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2027-03-24 (Estimated); Study Completion 2027-03-24 (Estimated)

PRIMARY OUTCOMES:
Pathologically confirmed progression free survival | 2 years
  To estimate pathologically confirmed progression free survival (pPFS) two years post-operatively in HPV associated OPC patients who undergo active surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Acharf Shamseddine, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Baptist Alliance MCI (Data Collection Only), Miami, Florida
  - Memorial Sloan Kettering Basking Ridge (Limited protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activites), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org